CLINICAL TRIAL: NCT02971501
Title: A Phase II Trial of Osimertinib (AZD9291) With or Without Bevacizumab in Patients With EGFR Mutation Positive NSCLC and Brain Metastases
Brief Title: Osimertinib With or Without Bevacizumab in Treating Patients With EGFR Positive Non-small Cell Lung Cancer and Brain Metastases
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01733; NCI-2016-01733 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2000021123; 10042; 10042 (Other: Yale University Cancer Center LAO); 10042 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Lung Non-Small Cell Carcinoma; Metastatic Malignant Neoplasm in the Brain; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms; Lung Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (osimertinib, bevacizumab) (Experimental): Patients receive osimertinib PO QD on days 1-21 and bevacizumab IV over 30-90 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, MRI, tumor biopsy and blood sample collection throughout the study.
  Interventions: Biological: Bevacizumab; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Osimertinib
- Arm II (osimertinib) (Experimental): Patients receive osimertinib PO QD on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, MRI, tumor biopsy and blood sample collection throughout the study.
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Arm I (osimertinib, bevacizumab)
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
  Arms: Arm I (osimertinib, bevacizumab)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Arm I (osimertinib, bevacizumab)
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
  Arms: Arm I (osimertinib, bevacizumab)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
  Arms: Arm I (osimertinib, bevacizumab)
Drug: Osimertinib — Given PO
  Other Names: AZD 9291; AZD-9291; AZD9291; Mereletinib

SUMMARY:
This phase II trial studies how well osimertinib with or without bevacizumab works in treating patients with EGFR positive non-small cell lung cancer that has spread to the brain (brain metastases). Osimertinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Bevacizumab may stop or slow non-small cell lung cancer by blocking the growth of new blood vessels necessary for tumor growth. Giving osimertinib with or without bevacizumab may work better in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the progression-free survival with osimertinib (AZD9291) plus bevacizumab compared to osimertinib (AZD9291) alone.

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of the combination of osimertinib (AZD9291) and bevacizumab.

II. To evaluate the time to progression in the central nervous system (CNS) with osimertinib (AZD9291) plus bevacizumab versus single-agent osimertinib (AZD9291).

III. To determine the overall response rate and the intracranial response rate to the combination versus single agent.

IV. To assess the overall survival in patients receiving osimertinib (AZD9291) plus bevacizumab compared to osimertinib (AZD9291) alone.

TRANSLATIONAL OBJECTIVES:

I. To investigate mechanisms of sensitivity and resistance to combination osimertinib (AZD9291) plus bevacizumab versus osimertinib (AZD9291) by molecularly characterizing tumor samples including T790M status.

II. To assess whether circulating tumor deoxyribonucleic acid (DNA) in plasma can be used as an indicator of sensitivity and resistance to treatment.

III. To determine whether an angiogenic signature using a multiplex panel array is associated with benefit from the combination of osimertinib (AZD9291) plus bevacizumab.

IV. To investigate angiogenesis, immune and signaling pathway markers in tumor samples to determine biomarkers predictive of benefit from combination therapy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive osimertinib orally (PO) once daily (QD) on days 1-21 and bevacizumab intravenously (IV) over 30-90 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive osimertinib PO QD on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients undergo computed tomography (CT) scan, magnetic resonance imaging (MRI), tumor biopsy and blood sample collection throughout the study.

After completion of study treatment, patients are followed up for a minimum of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer (NSCLC) with an activating EGFR mutation (exon 19 deletion, L858R point mutation, or any other mutation known to be associated with EGFR TKI sensitivity); presence of an activating EGFR mutation may be documented in tumor tissue or by plasma testing if performed in a Clinical Laboratory Improvement Act (CLIA)-certified laboratory
* No prior treatment with an EGFR TKI; patient may have received prior chemotherapy for early-stage or advanced disease but this is not required; prior immunotherapy is not allowed
* Patients must have at least one measurable CNS lesion that is asymptomatic, untreated, and does not require local therapy at the time of enrollment; measurable CNS disease is defined as a brain metastasis that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 5 mm (>= 0.5 cm) with brain magnetic resonance imaging (MRI); if the lesion is 5-10 mm in size and is the only measurable disease, MRI imaging must be performed with 1.5 mm slice thickness or less; a history of previously treated brain metastases is allowed, however any lesion present at the time of whole brain radiotherapy or included in the stereotactic radiotherapy field (or within 2 mm of the treated lesion) will NOT be considered "untreated" unless it is new or documented to have progressed unequivocally since treatment
* Patients are not required to have measurable systemic (i.e. non-CNS) disease; if present, measurable systemic disease must be able to be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) with conventional techniques or as >= 10 mm (>= 1 cm) with spiral computed tomography (CT) scan, MRI, or calipers by clinical exam
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Life expectancy of greater than 3 months
* The use of anti-convulsants is allowed, as long as the patient is on a stable dose with no seizure activity for at least 2 weeks prior to initiating trial therapy
* Female subjects should be using highly effective contraceptive measures, and must have a negative pregnancy test and not be breast-feeding prior to start of dosing if of child- bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

  * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
  * Women under 50 years old would be consider postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the post-menopausal range for the institution
  * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
* Fertile men should be willing to use barrier contraception during and for 4 months after osimertinib (AZD9291), and fertile women must agree to use adequate contraceptive measures during and for 6 weeks after osimertinib (AZD9291); fertile men and women must agree to use adequate contraceptive measures during study therapy and for at least 6 months after the completion of bevacizumab therapy; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the patient should inform the treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Symptomatic brain metastases or symptomatic leptomeningeal disease; asymptomatic leptomeningeal disease is allowed
* Patients with brain metastases for whom complete surgical resection is clinically appropriate
* Prior treatment with any EGFR TKI
* Prior treatment with agents targeting the VEGF pathway, including bevacizumab
* The use of corticosteroids to control cerebral edema or treat neurologic symptoms will not be allowed, and patients who previously required corticosteroids for symptom control must be off steroids for at least 3 days without recurrence of symptoms prior to starting trial therapy; corticosteroids for other indications is allowed
* Patients may not be receiving any other investigational agents and may not have participated in a study of an investigational agent or using an investigational device within five half-lives of the compound or 3 months, whichever is greater
* Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment with the exception of alopecia and grade 2 platinum-therapy related neuropathy
* Concurrent, active malignancies in addition to that being studied (other than cutaneous squamous cell carcinoma or basal cell carcinoma)
* Any contraindication to MRI (i.e. patients with pacemakers or other metal implanted medical devices)
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to osimertinib (AZD9291) or bevacizumab
* Urine protein should be screened by urine analysis; if protein is 2+ or higher, 24-hour urine protein should be obtained; patients with 24-hour urine protein >= 1000 mg are excluded
* Serious or non-healing wound, ulcer or bone fracture
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to day 1
* Invasive procedures defined as follows:

  * Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to day 1 therapy
  * Anticipation of need for major surgical procedures during the course of the study
  * Core biopsy within 7 days prior to day 1 (D1) therapy
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to day 1
* Patients with clinically significant cardiovascular disease are excluded

  * Inadequately controlled hypertension (HTN) (systolic blood pressure [SBP] > 160 mmHg and/or diastolic blood pressure [DBP] > 90 mmHg despite antihypertensive medication)
  * History of cerebrovascular accident (CVA) within 6 months (see additional requirement for adjuvant protocols)
  * Myocardial infarction or unstable angina within 6 months (see additional requirement for adjuvant protocols)
  * New York Heart Association grade II or greater congestive heart failure
  * Serious and inadequately controlled cardiac arrhythmia
  * Significant vascular disease (e.g. aortic aneurysm, history of aortic dissection)
  * Clinically significant peripheral vascular disease
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (Fridericia's correction formula [QTcF]) > 470 ms obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine derived corrected QT (QTc) value
  * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block, second degree heart block)
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval
* Evidence of bleeding diathesis or coagulopathy (including clinically significant hemoptysis)
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib (AZD9291)
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inducers of CYP3A4 (at least 3 weeks prior); all patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4
* Any evidence of severe or uncontrolled systemic diseases, including, but not limited to, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV); screening for chronic conditions is not required
* History of hypersensitivity active or inactive excipients of osimertinib (AZD9291) or drugs with a similar chemical structure or class to osimertinib (AZD9291)
* Absolute neutrophil count < 1.5 x 10^9/L
* Platelet count < 100 x 10^9/L
* Hemoglobin < 90 g/L
* Alanine aminotransferase > 2.5 times upper limit of normal (ULN) if no demonstrable liver metastases or > 5 times ULN in the presence of liver metastases; aspartate aminotransferase > 2.5 times ULN if no demonstrable liver metastases or > 5 times ULN in the presence of liver metastases
* Total bilirubin > 1.5 times ULN if no liver metastases or > 3 times ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia) or liver metastases
* Serum creatinine > 1.5 times ULN concurrent with creatinine clearance < 50 mL/min (measured or calculated by Cockcroft and Gault equation)-confirmation of creatinine clearance is only required when creatinine is > 1.5 times ULN
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From start of treatment to time of progression (in CNS or non-CNS disease) or death, whichever occurs first, assessed up to 5.5 years
  The two study arms will be compared for PFS with Kaplan-Meier estimates and log-rank tests. The Rothman confidence interval (CI) will be reported. In addition, the possible risk factors will be compared for survival with log-rank test. For multivariate analysis, the proportional hazards Cox model will be applied to investigate potential prognostic factors, such as age and stage of disease of the PFS data. The adjusted p-values of the hazard ratios and the adjusted 95% confidence interval will be reported.

SECONDARY OUTCOMES:
Overall survival (OS) | From start of treatment to death, assessed up to 5.5 years
  The two study arms will be compared for OS with Kaplan-Meier estimates and log-rank tests. The Rothman CI will be reported. In addition, the possible risk factors will be compared for survival with log-rank test. For multivariate analysis, the proportional hazards Cox model will be applied to investigate potential prognostic factors, such as age and stage of disease of the OS data. The adjusted p-values of the hazard ratios and the adjusted 95% confidence interval will be reported.
Incidence of adverse events | Up to 5.5 years
  Assessed by Common Terminology Criteria for Adverse Events. Adverse medical events will be tabulated. National Cancer Institute toxicity grade 1 to grade 4 laboratory abnormalities will be listed.
Overall response rate | Up to 5.5 years
  Will be estimated using the 95% confidence CI based on Wilson's method. The Wilcoxon rank sum test and Fisher's exact test will be applied to study the association between the response status and the continuous and categorical variables respectively.
Intracranial response rate | Up to 5.5 years
  Will be estimated using the 95% confidence CI based on Wilson's method. The Wilcoxon rank sum test and Fisher's exact test will be applied to study the association between the response status and the continuous and categorical variables respectively.
Time to intracranial progression | Up to 5.5 years
  Will be assessed by Response Assessment in Neuro-Oncology Brain Metastases.
Time to central nervous system (CNS) progression | From start of treatment to time of progression in the CNS, assessed up to 5.5 years
Objective response defined as a complete or partial response | Up to 5.5 years
  Will be determined by investigator assessment using Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1.

OTHER OUTCOMES:
Molecular characterization | Up to 2 years
  Analysis will be completed using Lasso-based elastic net method.
Circulating tumor deoxyribonucleic acid assessed in plasma | Up to 2 years
  Analysis will be completed using Lasso-based elastic net method.
Angiogenic signature assessed in plasma by multiplex panel array | Up to 2 years
  Analysis will be completed using Lasso-based elastic net method.
Biomarker analysis of angiogenesis and signaling pathways | Up to 2 years
  Analysis will be completed using Lasso-based elastic net method.
Changes in the tumor immune microenvironment | Baseline to 2 years
  Analysis will be completed using Lasso-based elastic net method.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah B Goldberg, Principal Investigator — Yale University Cancer Center LAO
Locations (18):
- United States (18):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Deng Z, Qin Y, Liu Y, Zhang Y, Lu Y. Role of Antiangiogenic Agents Combined With EGFR Tyrosine Kinase Inhibitors in Treatment-naive Lung Cancer: A Meta-Analysis. Clin Lung Cancer. 2021 Jan;22(1):e70-e83. doi: 10.1016/j.cllc.2020.08.005. Epub 2020 Sep 18. PMID 33067126